CLINICAL TRIAL: NCT01356498
Title: Multicenter, Open Label Extension Study of 8 mg PEG-uricase in Subjects Who Completed Protocols C0405 or C0406 for Symptomatic Gout
Brief Title: Open-Label Extension Study for Patients Who Completed a Phase 3 Double-blind Study of PEG-uricase for Symptomatic Gout
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Savient Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C0407
Record Dates: First submitted 2008-10-27; First posted 2011-05-19 (Estimated); Results first posted 2011-12-02 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-10

CONDITIONS: Gout
Keywords: gout; chronic gout
MeSH Terms: conditions — Gout | interventions — Pegloticase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- q2 RCT (Experimental): Pegloticase every 2 wk arm of Randomized Controlled Trial(RCT), continued to receive pegloticase every 2 weeks (q2 wk) or every 4 weeks (q4 wk) in Open Label Extention (OLE) study
  Interventions: Biological: pegloticase
- q4 RCT (Experimental): Pegloticase every 4 wk arm of Randomized Controlled Trial (RCT), continued to receive pegloticase every 2 weeks (q2 wk) or every 4 weeks (q4 wk) in Open Label Extention (OLE) study
  Interventions: Biological: pegloticase
- Placebo in RCT (Experimental): Placebo arm in Randomized Controlled Trial (RCT), received pegloticase every 2 weeks (q2 wk) or every 4 weeks (q4 wk) in OLE
  Interventions: Biological: pegloticase

INTERVENTIONS:
Biological: pegloticase — 8 mg intravenous infusion

SUMMARY:
This is an open-label extension phase of two double-blind, placebo-controled Phase 3 protocols evaluating PEG-uricase in the treatment of hyperuricemic subjects with symptomatic gout. The purpose of this study is to provide a continuation of treatment to subjects completing the double-blind studies and obtain long-term safety and efficacy data.

ELIGIBILITY:
Inclusion Criteria:

* Completed treatment in one of two double-blind, placebo controlled studies of PEG-uricase in subjects with hyperuricemia and symptomatic gout

Exclusion Criteria:

* unstable angina
* uncontrolled arrhythmia
* uncontrolled hypertension
* end stage renal disease requiring dialysis
* anemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2006-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, M.D., Study Director — Savient Pharmaceuticals, Inc.
Locations (22):
- United States (22):
  - Kaiser Permanente Medical Center, Clinical Trials Unit, San Francisco, California
  - Pacific Arthritis Center Medical Group, Santa Maria, California
  - Agilence Arthritis & Osteoporosis Medical Center, Whittier, California
  - Veterans Affairs Medical Center, Washington D.C., District of Columbia
  - Arthritis & Rheumatic Disease Specialties, Aventura, Florida
  - Ocala Rheumatology Research Center, Ocala, Florida
  - St. Petersburg Arthritis Center, St. Petersburg, Florida
  - The University of Chicago, Chicago, Illinois
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - Peter A. Holt, M.D., Baltimore, Maryland
  - Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Justus J. Fiechtner, MD, PC, Lansing, Michigan
  - CentraCare Clinic, Saint Cloud, Minnesota
  - Rheumatology Associates of North Jersey, Teaneck, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - New Horizons Clinical Research, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - STAT Research, Inc., Dayton, Ohio
  - David R. Mandel, MD, Inc., Mayfield Village, Ohio
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Mid Atlantic Research Assoc., Philadelphia, Pennsylvania
  - Arthritis Northwest, PLLC, Spokane, Washington

REFERENCES:
- [Derived] Pillinger MH, Fields TR, Yeo AE, Lipsky PE. Dissociation Between Clinical Benefit and Persistent Urate Lowering in Patients with Chronic Refractory Gout Treated with Pegloticase. J Rheumatol. 2020 Apr;47(4):605-612. doi: 10.3899/jrheum.190161. Epub 2019 Jun 15. PMID 31203212
- [Derived] Lipsky PE, Calabrese LH, Kavanaugh A, Sundy JS, Wright D, Wolfson M, Becker MA. Pegloticase immunogenicity: the relationship between efficacy and antibody development in patients treated for refractory chronic gout. Arthritis Res Ther. 2014 Mar 4;16(2):R60. doi: 10.1186/ar4497. PMID 24588936
- [Derived] Baraf HS, Becker MA, Gutierrez-Urena SR, Treadwell EL, Vazquez-Mellado J, Rehrig CD, Ottery FD, Sundy JS, Yood RA. Tophus burden reduction with pegloticase: results from phase 3 randomized trials and open-label extension in patients with chronic gout refractory to conventional therapy. Arthritis Res Ther. 2013 Sep 26;15(5):R137. doi: 10.1186/ar4318. PMID 24286509

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects completing one of the randomized, controlled Phase 3 clinical trials (RCTs) of pegloticase [C0405 and C0406 (NCT00325195)] were invited to participate in this open-label extension study.
Pre-assignment Details: Participants made the decision, along with the treating investigator, of which dose to receive in this study while remaining blinded to treatment received and results during the RCT. Cohort designations are based on participants' initial RCT treatment and whether uric acid remained <6 mg/dL for 80% of the time during months 3 and 6 in the RCT.
Groups:
- q2 RCT, Responder: Responder in Pegloticase every 2 wk arm of Randomized Controlled Trial (RCT), continued to receive pegloticase every 2 weeks (q2 wk) or every 4 weeks (q4 wk) in Open Label Extension (OLE) study
- q4 RCT, Responder: Responder in Pegloticase every 4 wk arm of Randomized Controlled Trial, continued to receive pegloticase every 2 weeks (q2 wk)or every 4 weeks (q4 wk)in Open Label Extension (OLE) study
- Placebo in RCT, q2 in OLE: Placebo arm in Randomized Controlled Trial (RCT), initiated pegloticase treatment every 2 weeks (q2 wk)in Open Label Extension (OLE) study
- q2 RCT, Non-responder: Non-responder in Pegloticase every 2 wk arm of Randomized Controlled Trial, continued to receive pegloticase every 2 weeks (q2 wk)or every 4 weeks (q4 wk)in Open Label Extension (OLE) study
- q4 RCT Non-responder: Non-responder in Pegloticase every 4 wk arm of Randomized Controlled Trial, continued to receive pegloticase every 2 weeks (q2 wk)or every 4 weeks (q4 wk)in Open Label Extension (OLE) study
- Placebo in RCT, q4 in OLE: Placebo arm in Randomized Controlled Trial (RCT), initiated pegloticase treatment every 4 weeks (q4 wk)in Open Label Extension (OLE) study
Period: Overall Study
Arm/Group | q2 RCT, Responder | q4 RCT, Responder | Placebo in RCT, q2 in OLE | q2 RCT, Non-responder | q4 RCT Non-responder | Placebo in RCT, q4 in OLE
Started | 35 | 25 (2 other patients received no investigational drug in C0407 but elected to be followed in Observation) | 23 | 22 | 28 | 16
Completed | 24 | 17 | 11 | 8 | 8 | 2
Not Completed | 11 | 8 | 12 | 14 | 20 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | q2 RCT, Responder | q4 RCT, Responder | Placebo in RCT, q2 in OLE | q2 RCT, Non-responder | q4 RCT Non-responder | Placebo in RCT, q4 in OLE | Total
Number analyzed (Participants) | 35 | 25 | 23 | 22 | 28 | 16 | 149
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 17 | 18 | 16 | 23 | 11 | 105
  >=65 years | 15 | 8 | 5 | 6 | 5 | 5 | 44
Age Continuous [Mean (Standard Deviation); unit: years] | 62.4 (13.66) | 58.6 (13.59) | 56.6 (10.53) | 52.0 (13.12) | 53.5 (12.25) | 54.6 (13.62) | 56.8 (13.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 7 | 4 | 4 | 4 | 3 | 32
  Male | 25 | 18 | 19 | 18 | 24 | 13 | 117
Region of Enrollment [Number; unit: participants]
  United States | 32 | 22 | 22 | 17 | 27 | 13 | 133
  Canada | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Mexico | 3 | 2 | 0 | 5 | 1 | 3 | 14

OUTCOME MEASURES:

1. Primary Outcome: Uric Acid (mg/dL)
Description: Uric acid measured at 3 month-intervals
Time Frame: Week 13, Week 25, Week 53, Week 101
Population: ITT
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | q2 RCT, Responder | q4 RCT, Responder | Placebo in RCT, q2 in OLE | q2 RCT, Non-responder | q4 RCT Non-responder | Placebo in RCT, q4 in OLE
Number analyzed (Participants) | 31 | 24 | 18 | 17 | 22 | 10
mg/dL
  OLE Week 13 | 1.33 (3.103) | 1.91 (4.082) | 5.06 (4.538) | 9.76 (1.346) | 9.66 (2.529) | 8.08 (3.561)
  OLE Week 25 | 1.4 (3.196) | 1.95 (3.761) | 4.69 (4.454) | 8.89 (3.984) | 9.94 (2.646) | 8.09 (3.536)
  OLE Week 53 | 0.87 (2.327) | 1.55 (3.690) | 2.7 (4.255) | 9.18 (2.946) | 9.59 (2.782) | 6.45 (3.248)
  OLE Week 101 | 0.84 (2.619) | 1.47 (3.317) | 4.29 (3.985) | 7.7 (4.244) | 9.42 (1.961) | 8.5 (NA) — One subject only

2. Secondary Outcome: Tophus Response
Description: Target tophi evaluated during the randomized, controlled study were followed for response at 3, 6, 12, 18 and 24 months in this open-label extention study. Results from each participant's final assessment on drug are reported (as last observation carried forward). Complete response=complete disappearance of at least one tophus with no new or worsening tophus. Partial Response=a 50% or more decrease in at least one tophus with no new or worsening tophus.
Time Frame: Up to 2 years
Population: ITT, Last observation(on drug) carried forward showing patients with an Overall Tophus Response of Complete or Partial Response.
Measure: Number; unit: participants
Arm/Group | q2 RCT, Responder | q4 RCT, Responder | Placebo in RCT, q2 in OLE | q2 RCT, Non-responder | q4 RCT Non-responder | Placebo in RCT, q4 in OLE
Number analyzed (Participants) | 23 | 14 | 16 | 16 | 20 | 5
participants
  Complete Response | 19 | 13 | 10 | 4 | 7 | 3
  Partial Response | 4 | 0 | 3 | 4 | 2 | 1

3. Secondary Outcome: Patient Reported Outcome: SF-36 Physical Component Summary Score
Description: SF-36 is the Medical Outcomes Survey Short Form-36, a 36-item self-reported questionnaire which assesses health-related limitations in 8 dimensions. The Physical Component Summary Score (PCS) is a composite summary score derived from the dimensions related to physical functioning outcomes: Physical Function, Role Physical, General Health and Bodily Pain (each with a 0 to 100 scale where 0=worst, 100=best).
  The Summary Score is constructed as a T-score with a mean of 50 and standard deviation of 10, where higher scores indicate a better health status.
Time Frame: RCT Week 25; OLE Week 25; OLE Week 53, OLE Week 77, OLE Week 101
Population: Number of participants was the subset of the ITT population with SF-36 baseline data
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- q2 RCT, Responder: Responder in Pegloticase every 2 wk arm of RCT, continued to received pegloticase (q2 wk or q4 wk) in OLE
- q4 RCT Responder: REsponder in Pegloticase every 4 wk arm of RCT, contuned to received pegloticase (q2 wk or q4 wk) in OLE
- Placebo in RCT, q2 in OLE: Placebo arm in RCT, initiated pegloticase treatment q2 wk in OLE
- q2 RCT, Non-responder: Non-responder in pegloticase every 2 wk arm of RCT, continued to received pegloticase (q2 wk or q4 wk) in OLE
- q4 RCT, Non-responder: Non-responder in Pegloticase every 4 wk arm of RCT, continued to received pegloticase (q2 wk or q4 wk) in OLE
- Placebo in RCT, q4 in OLE: Placebo arm in RCT, initiated pegloticase treatment q4 wk in OLE
Arm/Group | q2 RCT, Responder | q4 RCT Responder | Placebo in RCT, q2 in OLE | q2 RCT, Non-responder | q4 RCT, Non-responder | Placebo in RCT, q4 in OLE
Number analyzed (Participants) | 34 | 25 | 23 | 19 | 26 | 15
units on a scale
  Baseline value (pre-pegloticase) | 34.92 (10.988) | 34.11 (10.022) | 27.55 (11.405) | 33.71 (11.581) | 32.8 (10.129) | 36.2 (11.926)
  Final Visit value (LOCF) | 40.40 (13.393) | 40.82 (7.482) | 30.34 (11.132) | 37.68 (10.298) | 34.76 (11.413) | 38.8 (13.155)

4. Secondary Outcome: Gout Flare Frequency
Description: The the mean number of flares per subject (flare frequency)was assessed over 3-month periods for up to 2 years of treatment
Time Frame: Up to 2 years
Population: Analysis is based on ITT population, and is presented by intervals of time on pegloticase
Measure: Mean (Standard Deviation); unit: Flares
Arm/Group | q2 RCT, Responder | q4 RCT, Responder | Placebo in RCT, q2 in OLE | q2 RCT, Non-responder | q4 RCT Non-responder | Placebo in RCT, q4 in OLE
Number analyzed (Participants) | 35 | 25 | 23 | 22 | 28 | 16
Flares
  Months 1-3 | 0.4 (0.69) | 0.8 (0.90) | 2.3 (2.91) | 0.6 (0.90) | 1.3 (1.49) | 1.5 (1.41)
  Months 4-6 | 0.4 (0.96) | 0.7 (0.95) | 1.3 (2.17) | 1.0 (1.73) | 0.8 (0.94) | 0.8 (1.18)
  Months 7-9 | 0.0 (0.17) | 0.3 (0.54) | 1.2 (1.80) | 0.6 (1.20) | 0.6 (0.97) | 0.4 (1.01)
  Months 10-12 | 0.1 (0.30) | 0.2 (0.51) | 0.6 (1.18) | 0.9 (1.34) | 0.9 (1.46) | 0.4 (0.63)
  Months 16-18 | 0.1 (0.25) | .3 (0.44) | 0.2 (0.40) | 0.7 (1.18) | 0.6 (0.85) | 0.4 (0.89)
  Months 22-24 | 0.1 (0.37) | 0.1 (0.23) | 0.4 (0.67) | 0.3 (0.65) | 0.6 (0.53) | 0.7 (1.15)

5. Secondary Outcome: Gout Flare Incidence
Description: Percentage of participants remaining in the study during the specified interval who experienced a gout flare during this interval.
Time Frame: Assessed in 3-month intervals up to 2 years
Population: The flare incidence is reported as the percentage of participants reporting flares during each 3-month interval.
Measure: Number; unit: Percentage of participants
Arm/Group | q2 RCT, Responder | q4 RCT, Responder | Placebo in RCT, q2 in OLE | q2 RCT, Non-responder | q4 RCT Non-responder | Placebo in RCT, q4 in OLE
Number analyzed (Participants) | 35 | 25 | 23 | 22 | 28 | 16
Percentage of participants
  Months 1-3 | 25.7 | 56.0 | 65.2 | 45.5 | 67.9 | 68.8
  Months 4-6 | 23.5 | 40.0 | 45.0 | 35.0 | 50.0 | 38.5
  Months 7-9 | 3.0 | 24.0 | 43.8 | 27.8 | 42.9 | 22.2
  Months 10-12 | 9.4 | 16.7 | 28.6 | 47.1 | 45.0 | 28.6
  Months 16-18 | 6.5 | 25.0 | 18.2 | 33.3 | 38.9 | 20.0
  Months 22-24 | 3.4 | 5.3 | 27.3 | 25.0 | 55.6 | 33.3

ADVERSE EVENTS:
Time Frame: Up to 30 days post-treatment (maximum of 32 months)
Description: Serious Adverse Events are reported for subjects during the On-pegloticase period, and includes events reported through 30 days after the last exposure to pegloticase.
Arm/Group | q2 RCT, Responder | q4 RCT, Responder | Placebo in RCT, q2 in OLE | q2 RCT, Non-responder | q4 RCT Non-responder | Placebo in RCT, q4 in OLE
Serious Adverse Events (participants affected / at risk) | 9/35 | 7/25 | 8/23 | 7/22 | 12/28 | 8/16
Other Adverse Events (participants affected / at risk) | 34/35 | 25/25 | 23/23 | 21/22 | 28/28 | 15/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | q2 RCT, Responder (N=35) | q4 RCT, Responder (N=25) | Placebo in RCT, q2 in OLE (N=23) | q2 RCT, Non-responder (N=22) | q4 RCT Non-responder (N=28) | Placebo in RCT, q4 in OLE (N=16)
Infusion related reaction (General disorders) | 1 | 0 | 4 | 1 | 3 | 3
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 2 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Arthritis Bacterial (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urinary Tract Infection Bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Gout (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 1 | 1
Renal Failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 0
Renal Failure Chronic (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 1 | 0
Azotemia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Diverticular Performation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Peritonitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 2 | 0 | 1 | 0
Femoral Artery Occlusion (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 1 | 0 | 1 | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Intentional Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Carotid Artery Stenosis (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hepatic Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lumbar Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0
Fluid Overload (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Suicide Attempt (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Goitre (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myeloproliferative Disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin Necrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Inguinal Hernia Repair (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | q2 RCT, Responder (N=35) | q4 RCT, Responder (N=25) | Placebo in RCT, q2 in OLE (N=23) | q2 RCT, Non-responder (N=22) | q4 RCT Non-responder (N=28) | Placebo in RCT, q4 in OLE (N=16)
Gout (Musculoskeletal and connective tissue disorders) | 15 | 19 | 19 | 16 | 24 | 13 — Preferred Term 'Gout' includes the preferred term for lower level term 'gout flare'
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 7 | 6 | 1 | 8 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 5 | 8 | 4 | 1 | 6 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 4 | 9 | 3 | 3 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 0 | 3 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 4 | 1 | 0 | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 1 | 1 | 0
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 1 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 2 | 2 | 0
Upper Respiratory Tract Invection (Infections and infestations) | 8 | 8 | 4 | 3 | 4 | 0
Urinary Tract Infection (Infections and infestations) | 7 | 5 | 2 | 2 | 4 | 0
Nasopharyngitis (Infections and infestations) | 3 | 5 | 1 | 1 | 4 | 1
Sinusitits (Infections and infestations) | 4 | 2 | 1 | 5 | 3 | 0
Cellulitis (Infections and infestations) | 2 | 1 | 2 | 3 | 3 | 1
Bronchitis (Infections and infestations) | 6 | 0 | 2 | 0 | 2 | 1
Gastroenteritis Viral (Infections and infestations) | 1 | 2 | 3 | 3 | 1 | 0
Influenza (Infections and infestations) | 0 | 3 | 1 | 3 | 2 | 1
Localised Infection (Infections and infestations) | 2 | 1 | 3 | 0 | 1 | 0
Infusion Related Reaction (General disorders) | 7 | 6 | 13 | 8 | 19 | 12
Oedema Peripheral (General disorders) | 7 | 6 | 5 | 1 | 2 | 0
Fatigue (General disorders) | 7 | 3 | 5 | 0 | 0 | 0
Chest Pain (General disorders) | 1 | 1 | 2 | 2 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 7 | 6 | 3 | 2 | 4 | 0
Nausea (Gastrointestinal disorders) | 3 | 5 | 2 | 2 | 5 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3 | 1 | 2 | 3 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 3 | 1 | 2 | 1
Abdominal Pain (Gastrointestinal disorders) | 2 | 2 | 2 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 4 | 2 | 1 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3 | 2 | 1 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 3 | 2 | 0 | 0 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 2 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 3 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1 | 1 | 1
Headache (Nervous system disorders) | 4 | 5 | 4 | 2 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 3 | 0 | 2 | 1 | 0
Hypertension (Vascular disorders) | 3 | 2 | 3 | 3 | 1 | 0
Flushing (Vascular disorders) | 1 | 3 | 1 | 2 | 1 | 0
Hypotension (Vascular disorders) | 1 | 2 | 1 | 0 | 3 | 0
Cataract (Eye disorders) | 2 | 3 | 1 | 0 | 2 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 2 | 0 | 2 | 1 | 0 | 2
Haematuria (Renal and urinary disorders) | 2 | 1 | 1 | 1 | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1 | 1 | 3 | 1
Depression (Psychiatric disorders) | 1 | 1 | 1 | 1 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days